CLINICAL TRIAL: NCT02801721
Title: Long Term Effect of Early Iron Supplementation and Psychosocial Stimulation on Growth and Development of Iron-deficient Anaemic Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PR-15059
Record Dates: First submitted 2016-06-05; First posted 2016-06-16 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Anaemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stimulation (Active Comparator): Stimulation group received psycho social stimulation. In the stimulation there were anemic and non anemic children. All anemic children received iron(syrup) supplementation.
  Interventions: Other: psycho social stimulation
- No stimulation (No Intervention): No stimulation group did not receive any stimulation. In the no stimulation group there were anemic and non anemic children. All anemic children received iron (syrup) supplementation

INTERVENTIONS:
Other: psycho social stimulation — The psychosocial intervention lasted for 9 months and included play demonstrations at home by a play leader (PL) who was trained to visit homes and teach the mothers about child development and care practices. They also showed the mothers how to play with children using toys in a way to promote good child development. In the original study all anemic children in early childhood received 30 mg ferrous sulphate daily based on recommendations from both the WHO (2003) and IOM reports (2001) for 6 months.
  Arms: Stimulation

SUMMARY:
1. Burden: Anaemia is a public health problem in our country. Fifty one percent young children aged 6 to 59 months are suffering from anaemia in Bangladesh (BDHS-2011) and the main cause of this problem is iron deficiency. Research findings show that Iron deficiency leads to delayed development and even reduce working capacity. All these impact negatively on quality of life and loss of national gross domestic product (GDP).
2. Knowledge gap: Little is known about long-term effects of early life iron deficiency anemia on development and behaviour of children after correction with iron supplements. There is also scarcity of information if early life psychosocial stimulation added to iron supplementation to these anemic children have long term benefits compared to non-stimulated anaemic children or non-anaemic children
3. Relevance:

   The aim was to conduct a follow up study to examine whether the IDA children, who recovered from iron deficiency and received additional more intense psychosocial intervention catch up to their optimum development in later life at school age, similar like non-anaemic peers.
4. Hypothesis (if any):

   1. The benefit of early iron supplementation in addition to Psychosocial stimulation on growth and development of IDA infants appears in later life.
   2. Addition of early psychosocial stimulation in treated IDA children help them catch up to their non-anemic peers in development over time.
5. Study Objective(s)

   1. To determine the long term effect of early psychosocial stimulation provided at the age of 6-24 months in addition to iron treatment in IDA children on their growth (height, weight and Head Circumference), IQ, executive function, school achievement, fine motor, memory and behaviour
   2. To compare the growth and development of IDA infants with non-anemic infants after 7 years of an intervention with iron supplementation and psychosocial stimulation.
6. Methods:

Sample: All children who participated in the iron and stimulation study at the age of 6 to 24 months (n=424).

Identification of sample: Using the addresses and by tracking through available mobile phone numbers.

Measurements

In the current follow-up, at the age of around 8-9 years all the available children will be measured for:

* WASI: The Wechsler Abbreviated Scale of Intelligence - Second Edition (WASI-II)
* School achievement
* Number Stroop
* SDQ (strength and difficulties):The Strengths and Difficulties Questionnaire (SDQ)
* Memory test of NEPSY (neuropsychological test)
* Digit span forward and backward
* Middle childhood HOME
* Fine motor skills using the Purdue peg board or Movement Assessment Battery Children- 2 (age -band 2 for 7-10 years)
* SES Anthropometric measurement: Children's height, weight and head circumference

DETAILED DESCRIPTION:
Millions of young children in developing countries have developmental deficits due to some preventable factors like poor nutrition, lack of a stimulating environment, and poverty. Although Bangladesh is doing well in achieving MDGs, still poor nutrition, poverty and poor parental education are prevalent. These mutually exclusive factors have an implication not only for the individuals' future but also for national income and development.

Usually, iron deficiency in the neonatal period and early childhood is considered a key to the development of disturbances in cognitive development. There is increasing evidence that iron deficiency anemia detrimentally affects children's development. Many cross sectional studies have shown that iron deficiency is associated with poor psycho motor development and behavioral deficits in young children, and poor cognition and school achievement in school-aged children. However, anemia is associated with many adverse social and economic family circumstances which may adversely affect children's development.

Nutrition along with early child development interventions can have additive or synergistic effects on child development, and in some cases, nutritional outcomes. Meta analysis, studies conducted in low, middle and high income countries in randomized controlled trials among primary school aged children (5-12 years) showed that concurrent iron supplementation improved global cognitive scores and growth and reduced risk of anemia and iron deficiency among anemic children by 50% and 75% respectively. According to the Lancet reviews on child development iron deficiency anemia during early childhood, when brain growth spurt occurs is one of the identified risk factor for later development. Similarly early psycho social stimulation acts as a protective factor in optimizing later development. Studies in Indonesia and Canada both found benefits from iron treatment to infants' motor development but not to mental development. It has been suggested that the poor level of mental development found in IDA infants may be irreversible in some circumstances. One systematic review and meta analysis revealed that daily iron supplementation in 2 to 5 years children increases hemoglobin and ferretin but has limited evidence in cognitive development and physical growth..

Anemia is a public health problem in Bangladesh where 51% of young children aged 6 to 59 months are suffering and the main cause of this problem is iron deficiency. A study conducted in Bangladesh found a non significant benefit to motor development from iron alone however the power of the study was extremely limited and the group receiving iron and zinc benefited in motor development. We also conducted a cluster randomized controlled trial in 2007-2008 on 6-24 months old iron deficient anemic (IDA) and non- anemic non-iron deficient (NANI) children with iron supplementation to IDA children for 6 months and weekly psycho social stimulation to all children in the stimulation clusters for 9 months in Bangladesh. The result showed that although the intervened IDA group recovered from their iron deficient status after 9 months, hey had significantly lower psycho motor development index (PDI) and responsiveness to the examiner compared to NANI group. Random-effects multilevel regressions of the developmental scores showed that psycho social stimulation improved children's mental development Index (MDI) in both the group. Interaction between iron status and stimulation showed a suggestive trend indicating that children with IDA and NANI responded differently to stimulation, i.e. the IDA group improved less than the NANI group. During that time we predicted that benefit of Iron supplementation and psycho social stimulation on children may appear in later life with application of more sensitive measurement tools for intelligence. The present study provides us a unique opportunity to examine long term effect of early iron supplementation and psycho social stimulation on growth and development of iron deficient anemic children.

Hypothesis:

3. The benefit of early iron supplementation in addition to Psycho social stimulation on growth and development of IDA infants appears in later life.

4. Addition of early psycho social stimulation in treated IDA children help them catch up to their non-anemic peers in development over time.

Study Objective(s)

1. To determine the long term effect of early psycho social stimulation provided at the age of 6-24 months in addition to iron treatment in IDA children on their growth (height, weight and Head Circumference), IQ, executive function, school achievement, fine motor and behavior
2. To compare the growth and development of IDA infants with non-anemic infants after 7 years of an intervention with iron supplementation and psycho social stimulation.

Study Setting Location: 30 villages of Monohardi Upazilla under Narsingdi district. Study design: Follow-up of a cluster randomized controlled trial. In the original study randomization was done at village level for psycho social stimulation. Two hundred and twelve children (106 anemic and 106 non anemic) aged 6-12 months in the "stimulation-villages (S)" received age specific psycho social stimulation and 212 children of "non-stimulation villages (NS: 106 anemic and 106 non anemic) were enrolled as controls. Mild and moderately anemic (Hb 80.0-109 g/L) and iron deficient (ferritin <12 μg/L) children of all the assigned villages (both S and NS) received ferrous-sulphate (Fe2SO4) syrup. Children were considered non-anemic if they had Hb>110 g/L and ferritin levels ≥12 μg/L. For all groups parental education were less than X grade.

Sample: All children who participated in the original study at the age of 6 to 24 months and can be located will be enrolled.

IDA group: All the children who were identified as IDA during early childhood (6-24 months) based on Hb level between 80-110 g/L and sTfR levels ≥ 5.0 mg/L.

Non-anemic group: All the children who were identified as NANI during early childhood based on Hb >110g/L and sTfR <5.0 mg/L) living in the same rural areas. .

Identification of sample: the study will try to track the children through their addresses and available mobile phone numbers that are registered during their enrollment. The study will also contact the local staff who worked as the play leaders and health workers and had close contact with the families to help us locate the children.

Randomization: In the original study the villages with at least 12 children (6 IDA and 6 NANI) aged 6-24 months were selected and randomly assigned to either psycho social stimulation or non-stimulation groups.

Intervention In the original study all anemic children in early childhood received 30 mg ferrous sulfate daily based on recommendations from both the WHO and IOM reports for 6 months. The psycho social intervention lasted for 9 months and included play demonstrations at home by a play leader (PL) who was trained to visit homes and teach the mothers about child development and care practices. The study showed the mothers how to play with children using toys in a way to promote good child development.

Plan of work: After taking written consent, the identified mothers and children will be interviewed for home based measurements (SES, HOME & SDQ) by team of two members - one trained testers (graduates in psychology or social science) and one health worker (high school graduate). The mother will be invited to come along with their children to the test centers (centrally located in the village) for developmental and anthropocentric assessments. The same tester will conduct the psychological assessments of the children while the health worker will assist in bringing and testing them. The testers and health workers will be unaware about the intervention group (blinded). Four teams will start assessments at the same time in 4 villages and rotate to the next after completing one. it is assumed that the testers will complete assessment of 10-12 children in one village in approximately two and half days.

Measurements

In the current follow-up, at the age of around 8-9 years all the available children will be measured for:

• WASI: The Wechsler Abbreviated Scale of Intelligence - Second Edition (WASI-II), a revision of the WASI, provides a brief, reliable measure of cognitive ability for use in clinical, educational and research settings. It consists of four sub tests: Vocabulary, Block Design, Similarities and Matrix Reasoning. Scores of these sub tests lead to calculate performance IQ (PIQ), verbal IQ (VIQ) as well as a full scale IQ (FSIQ). The average reliability coefficients of the WASI subtest range from .87 to .92 for the overall children's sample (Guilford1954 and Nunnally 1978). WASI has been used by this group in Bangladesh previously and was culturally adapted before use. The adapted and translated version has been assessed for face validity before use and showed meaningful correlation with nutritional and socio-economic variables (Ali- personal communication).

Previous study conducted by us showed that cognitive testing of pictures, piloted the original test on 35 children in Gaibandha and 20 children in Dhaka, and re-ranked the items according to difficulty. The test retest reliability of the adapted tool ranged from 0.77 to 0.86 for different subscales.

* School achievement: Children's school achievement will be measured using a locally developed test based on the 'wide range achievement test (WRAT) that measures mathematics, reading, writing and comprehension abilities. In addition their grade level, number of grades repeated, attendance in school, age of enrolment at primary school, age of leaving school, preschool attendance etc. will also be measured. This test has been used by a member of our group in a previous intervention study in rural Bangladesh and was sensitive to changes in serum iodine. This adapted version of school achievement test showed good face validity before testing. It also showed high concurrent validity (r=0.71) with Wechsler Intelligence Scale for Children (WISC-IV) at 10 years and moderately high predictive validity (r=0.54) of Wechsler Preschool and Primary Scale of Intelligence (WPPSI) used at 5 years in our recently completed cohort study in Bangladesh (Tofail -personal communication). It also showed meaningful correlation with socio-economic variables, parental education and children's nutritional status.
* Number Stroop: The number Stroop measures executive function of the children. It is a psychological test for mental (selective attention) vitality and flexibility. It has been used in Bangladesh in another study in Gaibandha where it picked up intervention effects (Ali- personal communication). We also used a modified word and color stroop test in Matlab that showed reasonable concurrent validity (r> 0.45) with other cognitive measures and socio-demographic variables .We will conduct a pilot test for number stroop in this study to assess face validity and test -retest reliability before using.
* Strength and difficulties questionnaire (SDQ): will be used to identify behavioral and emotional problems of the children based on mother's report. It is a widely and internationally used brief behavioral screening instrument assessing child positive and negative attributes across 5 sub-scales: 1) Emotional Symptoms, 2) Conduct Problems, 3) Hyperactivity-Inattention, 4) Peer Problems, 5) Pro social Behavior. The SDQ has been extensively researched with various populations and has been translated into over 40 languages. Reliability was generally satisfactory when assessed by internal consistency: (mean Cronbach α: 0.73), cross-informant correlation (mean: 0.34), or retest stability after 4 to 6 months (mean: 0.62) . Our team used it in several studies in Bangladesh and showed meaningful correlation of the sub-scales with socio-economic variables. We used the parent's report of SDQ and it showed good face validity and a conceptually meaningful pattern of cross-scale correlations and the acceptable internal reliability estimates found for each subscale. At five years of age it picked up intervention effect of prenatal supplementation in our recent analysis.
* Memory sub tests of NEuro PSYchological (NEPSY) Assessment: is a comprehensive instrument designed to assess neuro psychological development and provide insights regarding academic, social, and behavioral difficulties in preschool and school-age children. We will use only the memory test of NEPSY. We have used this memory test in one of our recent rural study on school children. Although it has been used in Bangladesh earlier but we will pilot it on current population to modify and adapt it accordingly.
* Digit span: Digit span forward and backward will be used to measure memory and executive function of the children. It has been used as a part of Wechsler Intelligence Scale for Children (WISC-IV) on 10 years old children and currently being used in one study on rural population. It showed good face validity and test retest reliability after 7 days. We will also pilot it on our current study area on non-study children to modify and adapt it accordingly before use.
* HOME: the middle childhood version of home observation for measurement of environment will be used to assess quality of home stimulation. Overall inter-observer reliability for the middle childhood -HOME reported to be satisfactory. Percentage agreement for specific items in the EC-HOME ranged from 79-100% while Cohen's kappa values ranged from 0.45 to 1. Intraclass correlation for subscale scores were in the interval of 0.79 to 0.94. The intraclass correlation for the total scale was 0.92. It has been used in several studies of Bangladesh and showed moderately high concurrent validity with IQ measures (r> 0.5).
* Fine motor skills using the Purdue peg board or Movement Assessment Battery for Children- 2 (age -band 2 for 7-10 years): it was prefered to conduct MABC-2, but we will make decision after piloting both the tests. Correlations between MABC-2 test components ranged between 0.25 and 0.36 (indicating little overlap between subtests). Correlation scores range from 0.73 to 0.84 for component scores and are equal to 0.80 for total test score. The study conducted earlier by us MABC in Bangladesh in younger children and MABC-2 in 8-year old children. This time a pilot study will be done on our current study area on non-study children to modify and adapt it accordingly before use.
* Socio economic status (SES) will be measured using a standard questionnaire. Anthropometric measurement: Children's height, weight and had circumference will be measured using standard measures.All these measures were culturally adapted in Bangladesh and have been used previously by our group. All the instruments are ready to use but will be pre-tested in the community before using.

Reliabilities Inter-observer reliabilities will be assessed on all measurements before the study begins and during the study on 10% of all the measurements.

Sample Size In the original study the sample size was calculated as 212 children in each of the IDA and NANI group considering 5% level of significance, 80% power, an improvement of 0.5 SD in children's development, an ICC of 0.01, design effect of 1.5 and 25% drop outs. In the follow-up we will assess all the available children of those groups. In the original study the analysis showed that there was no effect of clustering. Therefore we do not need to account for the design effect and the sample size without design effect will be 64 in each group. Considering a drop out of 10%, we need to enrol 70 children in each group and we believe it is possible to track that many children in those villages to have sufficient power to conduct the study.

Data Analysis After coding, the data will be entered in to a personal computer using SPSS 11.5 software. We will the check for normality of the data. Log transformation will be done if any data is positively skewed. The characteristics of the tested and lost groups will be compared using 'student t test' or ANOVA for continuous variables and χ2 for categorical variables. Pearson's bivariate correlation will be conducted to explore associations between the age of the child and each developmental measure.

The sociodemographic characteristics and growth measures at baseline will be compared between the IDA and NANI groups as well as between the stimulated and unstimulated groups by using random effects ANOVA.

Finally, it will be fitted random-effects multilevel regression model to the intelligence scores and nutritional outcome scores by using intention-to-treat analyses. We will investigate the effects of the IDA/NANI groups and stimulated/ unstimulated groups and their interaction. In each regression analysis, the outcome will be final developmental score, and we will adjust for the relevant initial score, along with the selected covariates that are identified as con-founders.

Data Safety Monitoring Plan (DSMP) Study questionnaires will be recorded on paper forms, which will be kept in a secure facility under the responsibility of the Principal Investigator of this study. All questionnaires and data forms will be reviewed for inconsistencies and missing data points. Edited data will be entered in a personal computer using SPSS.

Ethical Assurance for Protection of Human rights

Approval of the Research and Ethical Review Committees of icddr,b will be collected.

Written informed consent of one of the parents will be obtained after thorough explanation of the purpose of the study, requirements of participation, study procedures, and the risks and benefits to the child. Another person will be acting as witness at the time of consent signing.

Measures will be taken to ensure strict confidentiality of the information obtained.

ELIGIBILITY:
Inclusion Criteria:

* All non anaemic children
* Anaemic children (Haemoglobin concentration .80g/L and ,110g/L) and
* Serum transferrin receptor concentration ≥ 5.0mg/L

Exclusion Criteria:

* Twin Baby
* Children with known hematological diseases
* Children with known chronic diseases
* Refused concent

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 349 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cognitive ability | single time point at follow up after an average of 6 years of the original study
  We will use The Wechsler Abbreviated Scale of Intelligence (WASI) for measuring the cognitive ability. It consists of four subtests: Vocabulary, Block Design, Similarities and Matrix Reasoning. Scores of these subtests lead to calculate performance IQ (PIQ), verbal IQ (VIQ) as well as a full scale IQ (FSIQ). FSIQ will measure the cognitive ability.

SECONDARY OUTCOMES:
School achievement | single time point at follow up after an average of 6 years of the original study
  Children's school achievement will be measured using a locally developed test based on the 'wide range achievement test (WRAT) that measures mathematics, reading, writing and comprehension abilities.
Number Stroop | single time point at follow up after an average of 6 years of the original study
  The number Stroop measures executive function of the children. It is a psychological test for mental (selective attention) vitality and flexibility
Strength and difficulties questionnaire (SDQ) | single time point at follow up after an average of 6 years of the original study
  SDQwill be used to identify behavioural and emotional problems of the children based on mother's report. It is a widely and internationally used brief behavioural screening instrument assessing child positive and negative attributes
Memory subtests of NEuroPSYchological (NEPSY) Assessment | single time point at follow up after an average of 6 years of the original study
  NEPSYis a comprehensive instrument designed to assess neuropsychological development and provide insights regarding academic, social, and behavioural difficulties in preschool and school-age children.
Digit span | single time point at follow up after an average of 6 years of the original study
  Digit span forward and backward will be used to measure memory and executive function of the children.
Home Observation for Measurement of Environment (HOME) | single time point at follow up after an average of 6 years of the original study
  the middle childhood version of home observation for measurement of environment will be used to assess quality of home stimulation
Fine motor skills | single time point at follow up after an average of 6 years of the original study
  Fine motor skills using the Movement Assessment Battery for Children- 2 (age -band 2 for 7-10 years):
Socio economic status (SES) | single time point at follow up after an average of 6 years of the original study
  SES were measured using a standard questionnaire. We measure education level, job satatus, age, income ect of the parents. we also measure asset of the family etc through SES questionnaire.
Children's Height | single time point at follow up after an average of 6 years of the original study
  Children's height were measure by World Health Organization (WHO) guide line
Children's Weight | single time point at follow up after an average of 6 years of the original study
  Children's weight were measure by World Health Organization (WHO) guide line
Children's MUAC | single time point at follow up after an average of 6 years of the original study
  Children's MUAC were measure by World Health Organization (WHO) guide line
Children's OFC | single time point at follow up after an average of 6 years of the original study
  Children's OFC were measure by World Health Organization (WHO) guide line
Mother's height | single time point at follow up after an average of 6 years of the original study
  Mother's height were measure by World Health Organization (WHO) guide line
Mother's weight | single time point at follow up after an average of 6 years of the original study
  Mother's weight were measure by World Health Organization (WHO) guide line
Mother's MUAC | single time point at follow up after an average of 6 years of the original study
  Mother's MUAC were measure by World Health Organization (WHO) guide line

IPD SHARING:
Plan to Share IPD: Yes
if required we will share data with our expert

REFERENCES:
- [Result] Bodnar LM, Cogswell ME, McDonald T. Have we forgotten the significance of postpartum iron deficiency? Am J Obstet Gynecol. 2005 Jul;193(1):36-44. doi: 10.1016/j.ajog.2004.12.009. PMID 16021056
- [Result] Benton D; ILSI Europe a.i.s.b.l. Micronutrient status, cognition and behavioral problems in childhood. Eur J Nutr. 2008 Aug;47 Suppl 3:38-50. doi: 10.1007/s00394-008-3004-9. PMID 18683028
- [Result] Black MM, Baqui AH, Zaman K, Ake Persson L, El Arifeen S, Le K, McNary SW, Parveen M, Hamadani JD, Black RE. Iron and zinc supplementation promote motor development and exploratory behavior among Bangladeshi infants. Am J Clin Nutr. 2004 Oct;80(4):903-10. doi: 10.1093/ajcn/80.4.903. PMID 15447897
- [Result] Bryan J, Osendarp S, Hughes D, Calvaresi E, Baghurst K, van Klinken JW. Nutrients for cognitive development in school-aged children. Nutr Rev. 2004 Aug;62(8):295-306. doi: 10.1111/j.1753-4887.2004.tb00055.x. PMID 15478684
- [Result] Friel JK, Aziz K, Andrews WL, Harding SV, Courage ML, Adams RJ. A double-masked, randomized control trial of iron supplementation in early infancy in healthy term breast-fed infants. J Pediatr. 2003 Nov;143(5):582-6. doi: 10.1067/S0022-3476(03)00301-9. PMID 14615726
- [Result] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Result] Grantham-McGregor SM, Lira PI, Ashworth A, Morris SS, Assuncao AM. The development of low birth weight term infants and the effects of the environment in northeast Brazil. J Pediatr. 1998 Apr;132(4):661-6. doi: 10.1016/s0022-3476(98)70357-9. PMID 9580767
- [Result] Huda SN, Grantham-McGregor SM, Rahman KM, Tomkins A. Biochemical hypothyroidism secondary to iodine deficiency is associated with poor school achievement and cognition in Bangladeshi children. J Nutr. 1999 May;129(5):980-7. doi: 10.1093/jn/129.5.980. PMID 10222389
- [Result] Huda SN, Grantham-McGregor SM, Tomkins A. Cognitive and motor functions of iodine-deficient but euthyroid children in Bangladesh do not benefit from iodized poppy seed oil (Lipiodol). J Nutr. 2001 Jan;131(1):72-7. doi: 10.1093/jn/131.1.72. PMID 11208941
- [Result] Lind T, Lonnerdal B, Stenlund H, Gamayanti IL, Ismail D, Seswandhana R, Persson LA. A community-based randomized controlled trial of iron and zinc supplementation in Indonesian infants: effects on growth and development. Am J Clin Nutr. 2004 Sep;80(3):729-36. doi: 10.1093/ajcn/80.3.729. PMID 15321815
- [Result] Lozoff B, Jimenez E, Wolf AW. Long-term developmental outcome of infants with iron deficiency. N Engl J Med. 1991 Sep 5;325(10):687-94. doi: 10.1056/NEJM199109053251004. PMID 1870641
- [Result] Low M, Farrell A, Biggs BA, Pasricha SR. Effects of daily iron supplementation in primary-school-aged children: systematic review and meta-analysis of randomized controlled trials. CMAJ. 2013 Nov 19;185(17):E791-802. doi: 10.1503/cmaj.130628. Epub 2013 Oct 15. PMID 24130243
- [Result] Ruel MT, Alderman H; Maternal and Child Nutrition Study Group. Nutrition-sensitive interventions and programmes: how can they help to accelerate progress in improving maternal and child nutrition? Lancet. 2013 Aug 10;382(9891):536-51. doi: 10.1016/S0140-6736(13)60843-0. Epub 2013 Jun 6. PMID 23746780
- [Result] Thompson J, Biggs BA, Pasricha SR. Effects of daily iron supplementation in 2- to 5-year-old children: systematic review and meta-analysis. Pediatrics. 2013 Apr;131(4):739-53. doi: 10.1542/peds.2012-2256. Epub 2013 Mar 11. PMID 23478873
- [Result] Tofail F, Hamadani JD, Mehrin F, Ridout DA, Huda SN, Grantham-McGregor SM. Psychosocial stimulation benefits development in nonanemic children but not in anemic, iron-deficient children. J Nutr. 2013 Jun;143(6):885-93. doi: 10.3945/jn.112.160473. Epub 2013 Apr 24. PMID 23616511
- [Result] Walker SP, Wachs TD, Grantham-McGregor S, Black MM, Nelson CA, Huffman SL, Baker-Henningham H, Chang SM, Hamadani JD, Lozoff B, Gardner JM, Powell CA, Rahman A, Richter L. Inequality in early childhood: risk and protective factors for early child development. Lancet. 2011 Oct 8;378(9799):1325-38. doi: 10.1016/S0140-6736(11)60555-2. Epub 2011 Sep 22. PMID 21944375
- [Derived] Hossain SJ, Tofail F, Mehrin SF, Hamadani JD. Six-Year Follow-up of Childhood Stimulation on Development of Children With and Without Anemia. Pediatrics. 2023 May 1;151(Suppl 2):e2023060221E. doi: 10.1542/peds.2023-060221E. PMID 37125884